CLINICAL TRIAL: NCT06215651
Title: A Phase II, Single-arm, Multicenter, Prospective Study of Cadonilimab and Lenvatinib for Conversion Therapy in Unresectable Hepatocellular Carcinoma
Brief Title: Cadonilimab and Lenvatinib for Conversion Therapy in Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K4948
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Cadonilimab and Lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab and lenvatinib (Experimental): the combination therapy of Cadonilimab and Lenvatinib for conversion treatment in unresectable hepatocellular carcinoma
  Interventions: Drug: Cadonilimab lenvatinib

INTERVENTIONS:
Drug: Cadonilimab lenvatinib — ±TACE/HAIC
  Other Names: AK104

SUMMARY:
This study is a single-arm, open-label, exploratory clinical trial designed to assess the effectiveness and safety of the combination therapy of Cadonilimab and Lenvatinib for conversion treatment in unresectable hepatocellular carcinoma. Eligible patients, meeting the inclusion criteria and providing informed consent, will undergo 3-4 cycles of Cadonilimab and Lenvatinib conversion therapy. A single imaging assessment will be conducted, and successfully converted patients will proceed to surgical treatment, with pathological evaluation of intraoperative specimens. Post-surgery, patients will choose an appropriate adjuvant treatment based on prior treatment benefits, disease baseline, and personal preferences.

Patients who do not successfully convert and experience disease progression will exit the study for alternative treatment. Those who do not successfully convert but do not exhibit disease progression will continue conversion treatment with Cadonilimab and Lenvatinib±TACE/HAIC, with tumor imaging assessments every 3 cycles. Successfully converted patients will undergo surgery, followed by the selection of an appropriate adjuvant treatment based on prior treatment benefits, disease baseline, and personal preferences.

Patients who do not successfully convert and experience disease progression will exit the study for alternative treatment. Those who do not successfully convert but do not exhibit disease progression will continue conversion treatment with Cadonilimab and Lenvatinib±TACE/HAIC until disease progression or intolerable toxicity occurs, with a maximum treatment duration of 2 years. Efficacy assessment will use mRECIST and RECIST v1.1 criteria, and safety evaluation will follow CTCAE 5.0 standards. Adverse events will be recorded throughout the study, with a period extending to 60 days after treatment completion for serious adverse events or those related to Enfortumab Vedotin, and in some cases extended to 90 days post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign a written informed consent form before enrollment. Age >18 and ≤75 years, both genders are eligible. Patients with histologically or pathologically confirmed hepatocellular carcinoma (HCC) or meeting the clinical diagnostic criteria for HCC according to the American Association for the Study of Liver Diseases (AASLD).

BCLC stage C without distant or lymphatic metastasis, or BCLC stage B ineligible for curative surgical treatment.

Presence of measurable lesions (according to RECIST 1.1 criteria, CT scan long diameter ≥10 mm for non-lymph node lesions, CT scan short diameter ≥15 mm for lymph node lesions).

No prior systemic anticancer therapy. No prior local treatment for target lesions, including TAE, TACE, TARE, surgery, ablation, PEI, or radiotherapy.

Child-Pugh score <7. ECOG PS score: 0-1. At least one untreated measurable lesion according to RECIST v1.1, or a measurable lesion with confirmed progression after local treatment (e.g., radiofrequency ablation, ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, arterial embolization, arterial chemoembolization, etc.) per mRECIST criteria.

Expected survival >12 weeks. Non-surgically sterilized or premenopausal female patients must use a medically approved contraceptive measure during the study treatment period and within 3 months after the end of the study treatment. Pregnancy tests for non-surgically sterilized premenopausal female patients must be negative within 7 days before study entry, and they must not be lactating. Non-surgically sterilized or fertile male patients must agree to use a medically approved contraceptive measure with their female partners during the study treatment period and within 3 months after the end of the study treatment.

Adequate organ function, excluding any blood component and growth factor use within 14 days:

Hematology: ANC ≥1.5×10^9/L, PLT ≥50×10^9/L, HGB ≥90g/L. Liver function: TBIL ≤3×ULN, ALT and AST ≤5×ULN, serum albumin ≥28 g/L, ALP ≤5×ULN, and must be stable for at least 1 week after routine liver protection treatment as assessed by the investigator.

Renal function: Cr ≤1.5×ULN or creatinine clearance ≥50 mL/min (using the standard Cockcroft-Gault formula), and urine protein <2+; for patients with baseline urine protein ≥2+, a 24-hour urine collection and quantitative measurement with <1g of protein is required.

Coagulation function: INR and APTT ≤1.5×ULN; for subjects receiving anticoagulant therapy, PT and INR should be within the planned range.

Exclusion Criteria:

* Previously histologically/cytologically confirmed hepatocellular carcinoma with fibrolamellar components, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc.

Prior local or systemic anti-tumor therapy. History of hepatic encephalopathy. History of liver transplantation. Clinically significant pericardial effusion requiring drainage or clinically symptomatic pleural effusion.

Clinically evident ascites defined as detectable on physical examination or requiring drainage during screening.

Concurrent HBV and HCV infection (HCV RNA negative patients with a history of HCV infection are considered uninfected).

Central nervous system metastasis or leptomeningeal metastasis. History of esophageal or gastric variceal bleeding due to portal hypertension in the first 6 months before the initial dose. Participants must have undergone esophagogastroduodenoscopy within 6 months before the first dose; participants with severe (Grade 3) varices are not allowed to participate in the study.

Patients with any bleeding diathesis signs or history, experiencing any bleeding or hemorrhagic events ≥CTCAE Grade 3 within the first 4 weeks before the initial dose.

Occurrence of arterial or venous thromboembolic events in the first 6 months before the initial dose, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any severe history of thromboembolism. Exclusion criteria do not apply to stable thrombosis after routine anticoagulation therapy for implanted venous infusion ports or catheter-related thrombosis.

Uncontrolled hypertension, with systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg after optimal medical treatment, hypertensive crisis, or a history of hypertensive encephalopathy.

Symptomatic congestive heart failure (New York Heart Association Class II-IV) or echocardiographic left ventricular ejection fraction (EF) <50%. Symptomatic or poorly controlled arrhythmias, including atrial fibrillation or flutter with a ventricular rate >100 beats/min, a history of congenital long QT syndrome, or a corrected QT interval (QTc) >450 ms (male) or QTc >470 ms (female) on screening (using the Fridericia method). A history of myocarditis, cardiomyopathy, or malignant arrhythmias.

Severe bleeding tendency or coagulation disorders, or receiving thrombolytic therapy. Currently using or recently used (within 10 days before the first dose of study treatment) aspirin (>325 mg/day) or anticoagulants requiring INR monitoring (such as warfarin).

History of gastrointestinal perforation and/or fistula within the first 6 months before the initial dose, history of bowel obstruction (including incomplete bowel obstruction requiring parenteral nutrition), extensive colon resection (partial colon resection or extensive small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea.

Received radiation therapy within the first 3 weeks before the initial dose. Patients who received radiation therapy more than 7 days before the first dose can be enrolled. Presence of interstitial lung disease or interstitial lung disease requiring steroid treatment, either past or current.

Active pulmonary tuberculosis (TB), receiving anti-TB treatment, or having received anti-TB treatment within the past 1 year before the initial dose.

Subjects with any active autoimmune disease or a history of autoimmune disease (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, and those who have undergone thyroid surgery cannot be included). Subjects with resolved childhood asthma without the need for intervention can be included; subjects with asthma requiring bronchodilators for medical intervention cannot be included.

Subjects using immunosuppressive agents, either systemic or locally absorbable steroids for immunosuppressive purposes (dose >10 mg/day prednisone or equivalent), and still continuing within the last 2 weeks before enrollment.

Subjects with active infection or unexplained fever >38.5°C during screening or within the first 4 weeks before the initial dose (subjects with fever related to tumor-induced fever can be included according to the investigator's judgment).

Patients with objective evidence of past or present lung fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, or severe impairment of lung function.

Subjects with congenital or acquired immunodeficiency, such as HIV infection. Subjects who have not received live vaccines within 4 weeks before the study medication or may receive live vaccines during the study period.

Subjects with a known history of substance abuse, alcohol abuse, or drug abuse. Patients unable to take oral medication. The investigator deems it necessary to exclude subjects from this study. For instance, based on the investigator's judgment, if a participant has other factors that could potentially lead to the premature termination of the study, such as the presence of other serious illnesses (including mental disorders) requiring concurrent treatment, severe gastroesophageal varices, significant laboratory abnormalities, or factors related to family or social circumstances that could impact the safety of the participant or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Baseline up to approximately 6 months
  The proportion of patients whose tumor volume shrinks to a predetermined value and can maintain the minimum required duration, including complete response and partial response.
Conversion success rate | Baseline up to approximately 6 months
  Successful conversion criteria are as follows
  * Child-Pugh score <7
  * ECOG PS 0 or 1
  * No extrahepatic lesions or complete necrosis of extrahepatic lesions
  * Preservation of the intact vascular architecture of the liver
  * Adequate FLR after resection (≥35%)

SECONDARY OUTCOMES:
Disease control rate | Baseline up to approximately 6 months
  It refers to the proportion of patients whose tumor volume control (shrinkage or enlargement) reaches a predetermined value and can maintain the minimum required duration. According to the RECIST criteria (version 1.1), during the treatment period or within 30 days after the discontinuation of the investigational drug, it is the sum of the percentage of subjects who achieve complete response (CR), partial response (PR), and stable disease (SD).
Progression-free survival | Baseline up to approximately 12 months
  It refers to the time from the first administration of the regimen to the first occurrence of disease progression or death due to any cause in the subjects.
Overall survival | Baseline up to approximately 24 months
  The time from randomization to death due to any cause in the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Hai-Tao Zhao, Beijing, Beijing Municipality, China